CLINICAL TRIAL: NCT01301534
Title: Comparison of Methods to Improve Abdominal Aortic Aneurysm (AAA) Screening Rates in the Primary Care Setting.
Status: Completed | Type: Observational
Sponsor: Mike O'Callaghan Military Hospital (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: FWH20110041H
Record Dates: First submitted 2011-02-18; First posted 2011-02-23 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: abdominal aortic aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- T-Con: 1. Nurse initiated Telephone Consult (T-Con)
- Mail-Out: 2. Mail-0ut Letter to the patient
- Education: 3. Provider, Nurse and Technician Education with point-of-care patient referrals , Exam Room Flyer
- Control group: 4. Control group (i.e. usual care)

SUMMARY:
Standard of care dictates that eligible patients should receive an abdominal aortic aneurysm (AAA) screening ultrasound. At present, different military primary care physicians utilize different methods at their discretion to ensure their patients get screened-telephone contact; mail-out reminders; referring patients for ultrasound directly from an office visit; as well as other methods-which we will refer to as "usual care". The purpose of this study is to improve screening rates for AAA and determine what notification methods are best at improving screening rates.

DETAILED DESCRIPTION:
Approximately 1700 male patients (DoD beneficiaries) between the ages of 65-75 will be selected from their medical records. The information on the attached abstracted data sheet will be collected. As part of standard patient care operations, the Family Medicine and Internal Medicine Departments will inform patients on the need to receive a AAA screening ultrasound, based on their primary care manager's (PCM) preference for clinical notification:

1. Nurse initiated Telephone Consult (T-Con) (see attached)
2. Mail-0ut Letter to the patient (see attached)
3. Provider, Nurse and Technician Education with point-of-care patient referrals , Exam Room Flyer
4. Control group (i.e. usual care)

The Provider, Nurse and Technician Education will consist of a presentation given by the Principal Investigator (see attached PowerPoint) to the Family Medicine and Internal Medicine clinic staff and the posting of Exam Room Flyers in each Family Medicine and Internal Medicine exam room to prompt and encourage patient referrals for a AAA screening ultrasound.

Information requested on the attached abstracted data sheet will be used for initial identification of patients that should have a AAA screening ultrasound and again 3-4 months later to see if these same individuals received the procedure. All informational data sets will be totally de-identified by the Research Coordinator, Nellis Air Force Base, prior to releasing to the Principle Investigator.

The data will then be analyzed by Dr. Anneke Bush (WHMC statistician) and the results will be provided to the Principal Investigator for analysis.

ELIGIBILITY:
Inclusion:

* Tricare Insurance Beneficiary (military insurance) receiving care at Nellis AFB
* Male patients (DoD beneficiaries) between the ages of 65-75 years old.

Exclusion:

* Female patients.
* Non-English speaking.
* Patients who have already had abdominal CT scan, abdominal MRI, aortography or aortic ultrasound.
* Patients already diagnosed with AAA

Ages: 65 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: We will recruit approximately 1700 males (DoD beneficiaries) between the ages of 65-75 from their existing medical diagnostic records. There will be no special populations included. Some respondents may be patients of the PI however; the data sets received by the PI will be anonymous and will not be linked directly to the subjects.
Sampling Method: Non-Probability Sample
Enrollment: 1700 (Actual)
Dates: Start 2010-12; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
improving screening rates for AAA | 1 year
  Will the concerted use of (1) a nurse-initiated telephone consult (T-Con), (2) mail out reminder or (3) provider, nurse and technician education with point-of-care reminders be more successful than usual care at improving screening rates for AAA?

CONTACTS AND LOCATIONS:
Overall Officials: Ethan Zimmerman, M.D., Principal Investigator — Michael O'Callaghan Federal Hospital/Nellis Air Force Base
Locations (1):
- Michael O'Callaghan Federal Hospital/Nellis Air Force Base, Nellis Air Force Base, Nevada, United States